CLINICAL TRIAL: NCT05600504
Title: A Prediction Model for Early Prediction of Depression and Anxiety in Perioperative Elderly Adults
Brief Title: Development and Validation of a Prediction Model for Depression and Anxiety in Perioperative Elderly Adults
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Peking University First Hospital (Other); Peking University People's Hospital (Other); Shanghai Zhongshan Hospital (Other); Fudan University (Other); First Affiliated Hospital of Guangxi Medical University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Taihe Hospital (Other); Capital Medical University (Other); Beijing Tiantan Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); First Affiliated Hospital of Xinjiang Medical University (Other); China-Japan Friendship Hospital (Other); Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-DA-001
Record Dates: First submitted 2022-10-27; First posted 2022-10-31 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Predictive Model
Keywords: predicted model; depression; anxiety; elderly patient
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No depression: no intervention
  Interventions: Other: no intervention
- Depression: no intervention
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Anxiety and depression in later life are highly prevalent, often appear as comorbid disorders, and have many adverse consequences for both the individual and society. Given the disease burden, the large influx of new cases, and the economic costs, efforts should be made to prevent the onset of anxiety and depression in later life. Preventive interventions are likely to become more cost effective when they are targeted at elderly who have been exposed to risk factors known to be predictive of the onset of anxiety and/or depression. As the population aging is speeding up, senile diseases have become a significant and severe public health problem, influencing national health. More than 20 million elderly patients undergo surgery each year in China, accounting for a quarter of the population who undergo surgery. Therefore, it is necessary to construct a predictive model of anxiety and depression in perioperative elderly hospitalized patients

DETAILED DESCRIPTION:
More than 20 million elderly patients undergo surgery each year in China, accounting for a quarter of the population who undergo surgery. Therefore, it is necessary to construct a predictive model of anxiety and depression in perioperative elderly hospitalized patients. In 2015, the WHO introduced the concept of "healthy ageing" for global ageing, with a focus on the mental health of older people at its core.

Previous studies have found a 31 percent risk of anxiety and 29 percent risk of depression in older perioperative patients. Therefore, optimizing perioperative mental health management in older patients remains one of the challenges facing clinicians.

ELIGIBILITY:
Inclusion Criteria:

1. elective non-cardiac surgery,
2. American society of Aneshesiologists (ASA) classification Ⅰ ~ Ⅲ,
3. patients over age 65.

Exclusion Criteria:

1. patient refused follow-up study,
2. missing data exceeding 20%,
3. went to ICU or died after surgery,
4. have a history of any mental disorders such as epilepsy, Parkinson's disease, depression, anxiety, sleep disorders, or are currently taking relevant intervention drugs 5) patients with severe deafness, dementia or speech impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients, aged 65 years and above, who underwent elective non-cardiac surgeries in China during the period spanning from April 1, 2020, to April 30, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 6386 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Depression | Depression within 7 days of surgery
  Primary outcomes were depression Patient Health Questionnaire 9 (PHQ-9).The PHQ-9 is a nine-item questionnaire for screening on the presence of depressive symptoms and monitoring depression severity. Items were scored on a four-point scale with total scores ranging from zero to twenty-seven. Scores were defined as: ≥5 mild, ≥10 moderate, and ≥15 severe level of depression. The recommended screening cutoff was ≥10, corresponding with at least a moderate level of depression. The higher the score, the worse the situation. The total score ranges from 0 to 27, and higher scores indicate more depressive symptoms.

SECONDARY OUTCOMES:
Anxiety | Anxiety within 7 days of surgery
  The GAD-7 is a seven-item questionnaire for screening on the presence of generalized anxiety disorder and assessing its severity. Items were scored on a four-point scale with total scores ranging from zero to twenty-one. Scores were defined as: ≥5 mild, ≥10 moderate, and ≥15 severe anxiety. The recommended screening cutoff was ≥10, corresponding with at least a moderate level of anxiety. Higher scores mean more anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, PhD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided